CLINICAL TRIAL: NCT03775538
Title: A Randomised, Double-Blind, Multi-centre, Active Treatment, Extension and Safety Study for Patients With Idiopathic Parkinson's Disease (PD) Who Previously Completed the CDNF/DDS Main Study HP-CD-CL-2002
Brief Title: Safety of CDNF by Brain Infusion in Patients With Parkinson's Disease. Extension to HP-CD-CL-2002 Clinical Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Herantis Pharma Plc. (Industry)
Collaborators: Renishaw plc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-CD-CL-2003
Record Dates: First submitted 2018-10-11; First posted 2018-12-14 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease; Movement Disorders; Neuro-Degenerative Disease; Nervous System Diseases; Brain Diseases
Keywords: Parkinson; CDNF; Drug Delivery System; Intracerebral
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Nervous System Diseases; Brain Diseases

STUDY DESIGN:
Intervention Model Description: Randomised, Double-Blind, Active Treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDNF mid-dose (400 micrograms) (Experimental): Patients randomized to this group will receive 6 monthly-intermittent intracerebral doses of Cerebral Dopamine Neurotrophic Factor (CDNF) titrated to mid-dose (400 micrograms) administered via the Renishaw Drug Delivery System (DDS) to the bilateral putamen.
  Interventions: Drug: Cerebral Dopamine Neurotrophic Factor; Device: Renishaw Drug Delivery System
- CDNF high-dose (1200 micrograms) (Experimental): Patients randomized to this group will receive 6 monthly-intermittent intracerebral doses of Cerebral Dopamine Neurotrophic Factor (CDNF) titrated to high-dose (1200 micrograms) administered via the Renishaw Drug Delivery System (DDS) to the bilateral putamen.
  Interventions: Drug: Cerebral Dopamine Neurotrophic Factor; Device: Renishaw Drug Delivery System

INTERVENTIONS:
Drug: Cerebral Dopamine Neurotrophic Factor — Repeated intracerebral infusions
  Other Names: CDNF
Device: Renishaw Drug Delivery System — Stereotactically implanted device
  Other Names: DDS

SUMMARY:
This study is an extension to the HP-CD-CL-2002 clinical study. It evaluates the long-term safety and tolerability of CDNF in patients with Parkinson's disease when dosed directly into the brain using an implanted investigational drug delivery system (DDS). Long-term safety of the DDS is also being evaluated. All patients will receive monthly infusions of either mid- or high-dose of CDNF for a period of 6 months.

DETAILED DESCRIPTION:
A patient's participation in the study will last for six months and will include nine visits:

Screening (1 visit, same as HP-CD-CL-2002 End-of-Study visit) Dosing visits: CDNF (6 visits) DAT-PET (1 visit) End-of-study visit (1 visit)

Study examinations and assessments

* Physical examination: pulse rate, blood pressure, temperature, body weight and height, body mass index (BMI), neurological exam
* ECG (electrocardiography) and blood and urine tests
* Pregnancy tests for women of childbearing age
* Completion of a patient diary to record mobility and time asleep
* Parkinson's Kinetigraph (PKGTM) Data Logger: a watch-type movement recording device
* Questionnaires, rating scales and forms: quality of life, mood, memory, impulse control, mental health
* Assessment of the port and the skin around the port
* Cerebrospinal fluid sampling by lumbar puncture
* Magnetic resonance imaging (MRI)
* Positron emission tomography scans (PET)

For more information: https://treater.eu/clinical-study/

ELIGIBILITY:
Inclusion Criteria:

1. Completion of 6 months treatment period in the Main study (HP-CD-CL-2002) including End-of-Study assessment
2. Negative pregnancy test at study entry for females of childbearing potential. Willingness of using a highly effective form of contraception until 30 days after end of study. Males: willingness to use condom and not to donate sperm for 3 months following DAT-PET. Willingness of female partners of male study participants to use highly effective form of contraception until 30 days after their male partner's end of the study.
3. At least one functioning catheter in each putamen
4. Provision of informed consent

Exclusion Criteria:

1. Drug-resistant rest tremor, severe dyskinesia or severe head tremor, which could interfere with treatment infusions
2. Significant neurological disorder other than PD including clinically significant head trauma, cerebrovascular disease, epilepsy, CSF shunt or other implanted central nervous system device
3. Changes in pathology which give rise to safety concern such as sequelae from catheter implantation, clinically significant intracerebral trauma, oedema, haemorrhage, or infection
4. Current psychosis requiring therapy
5. Presence of clinically significant impulse control disorder by a positive screen on the QUIP-RS questionnaire score >20, or, presence of dopamine dysregulation syndrome
6. An unresolved intolerable adverse event or adverse device event in study HP-CD-CL-2002, which is not expected to resolve or cease to an acceptable level of intensity within reasonable time
7. Medical conditions, which might impair outcome measure assessments or safety measures
8. Impaired renal function
9. Concomitant treatment with neuroleptics or antipsychotic medication prescribed for treatment of current psychosis, central dopamine blockers or tricyclic antidepressants

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs)[safety-tolerability] | Week 40 to Week 65
  Total number, causality and severity of adverse events at any time during the study period
Change in Electrocardiogram (ECG): Ventricular rate, PR interval, qRS duration, QT, QTc [safety-tolerability] | Week 40, Week 53 and Week 65
  Changes in electrical activity of heartbeat measured by electrocardiogram: Ventricular rate (bpm), PR interval (msec), QRS duration (msec), QT (msec), QTc (msec)
Change in Beck Depression Inventory (BDI) score [safety-tolerability] | Week 40, Week 53 and Week 65
  Assessment of change in depression using Beck Depression Inventory (BDI) score: Sadness: Pessimism; Past Failure; Loss of pleasure; Guilty feelings; Punishment Feelings; Self-dislike; Self-criticalness;Suicidal thoughts or wishes; Crying; Agitation; Loss of interest; Indecisiveness;Worthlessness; Loss of energy; Changes in sleeping pattern; Irritability; Changes in appetite; Concentration difficulty; Tiredness or fatique; Loss of interest in sex. Rated on a 4-point scale ranging from 0 to 3 based on severity of each item (0=low intensity; 3=highest intensity). The maximum total score is 63.
Change in Questionnaire for impulsive-compulsive disorder in Parkinson's disease rating scale (QUIP_RS) [safety-tolerability] | Week 40, Week 53 and Week 65
  Assessment of changes in impulsive-compulsive disorders using QUIP_RS. Questions scored 0-4 (0=never; 4=very often) on gambling, sex, buying, eating, performing tasks/hobbies, repeating simple activities, and taking Parkinson's disease medication. Total QUIP-RS Score 0-112
Change in Montreal cognitive assessment (MoCA) [safety-tolerability] | Week 40, Week 53 and Week 65
  Assessment of change in cognitive domains using MoCA test: attention and, concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.
Changes in physical examination: anatomic findings [safety-tolerability] | Week 40 and Week 65
  Changes in anatomic findings found in physical examination of the following body systems: general inspection/upper extremities; head, eyes, ears, nose, throat, and superficial cervial lymph notes; neck, shoulders, back; chest and lungs; cardiovascular; abdomen; lower extremities
Changes in physical examination: clinical standard neurological examination | Week 40 and Week 65
  A clinical standard neurological examination by study investigator. Changes in motor function, sensory function, cranial nerve function (visual fields), cortical functions and reflexes are followed in the examination, scored as normal - abnormal without clinical relevance - abnormal with clinical relevance
Changes in vital signs: blood pressure [safety-tolerability] | Weeks 41, 45, 49, 53, 57, 61, and 63
  Changes in blood pressure during the study , measured as systolic and diastolic blood pressure (in mmHg)
Changes in vital signs: pulse rate [safety-tolerability] | Weeks 41, 45, 49, 53, 57, 61, and 63
  Changes in pulse rate during the study (in beats per minute)
Changes in vital signs: body temperature [safety-tolerability] | Weeks 41, 45, 49, 53, 57, 61, and 63
  Changes in body temperature during the study (in degrees celsius)
Changes in vital signs: body weight [safety-tolerability] | Weeks 41, 45, 49, 53, 57, 61, and 63
  Changes in body weight during the study (in kilograms)
Changes in vital signs: body mass index (BMI) [safety-tolerability] | Weeks 41, 45, 49, 53, 57, 61, and 63
  Changes in body mass index during the study (in kg/m^2)
Changes in clinical laboratory safety screen: clinical chemistry [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for clinical chemistry (Na, K, Urea, creatinine, creatine kinase, Ca, Bilirubin, IgG, Albumin, ALP, ALT, AST)
Changes in clinical laboratory safety screen: haematology - hemoglobin [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: hemoglobin (g/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: haematology - hematocrit [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: hematocrit (%, ratio of red blood cell volume to total blood volume). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: haematology - red blood cell (RBC) count [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: RBC count (10E12/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: mean cell volume (MCV) of red blood cells [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: MCV of red blood cells (fL). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: mean cell hemoglobin of RBC (MHC) [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: MCH (pg). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: Platelet count [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: Platelet count (10E9/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: white blood cell (WBC) counts [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: Cell counts (10E9/L) for total WBC, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: activated partial thromboplastin time (aPTT) [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: aPTT (sec) . Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: International Normalized Ratio (INR) [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for haematology: INR (standardized prothrombin time) to determine the effects of oral anticoagulants on the clotting system. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Changes in clinical laboratory safety screen: urinanalysis [safety-tolerability] | Weeks 40, 41, 45, 49, 53, 57, 61, and 65
  Changes in laboratory variables for urinanalysis (blood/erythrocytes, glucose, ketones, leukocytes, nitrites, pH, protein) studied by dipstick and scored 0-3. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance".
Formation of anti-CDNF antibodies [safety-tolerability] | Weeks 40, 45, 49, 53, 57, 61, and 65
  Formation and change in anti-CDNF antibody concentration (in ng/ml).
Device related occurrence of adverse device effects [safety-tolerability] | Week 40 to Week 65
  Occurrence of adverse device effects (ADE) at any time of the study period, for either the whole system or the individual sub systems (guide tubes/catheters, subcutaneous components, port), serious adverse device effect (SADE) including long term effects, neurological deficit (seizures), infection (local to components, in CNS), severe skin breakdown or necrosis requiring component removal life threatening or major (requiring intervention) intracerebral haemorrhage.

SECONDARY OUTCOMES:
Change in UPDRS (Unified Parkinson's Disease Rating Scale) Part III motor score [efficacy] | Week 40, Week 53 and Week 65
  Changes in severity of PD (Parkinson's disease) motor symptoms assessed by UPDRS Part III motor scores (each scored 0-4; 0=none, 4=severe): Speech; facial expression; tremor a rest; Tremor of hands; rigidity; firger taps; hand movelents; alternating movement of hands; leg agility; rising from chair; posture; gait; postural stability; body bradykinesia and hypokinesia. The total score, the sum of scores received from 27 assessments, is 0 - 108
Change in TUG (Timed Up and Go) test [efficacy] | Week 40, Week 53 and Week 65
  Changes in mobility assessed by TUG test (in minutes and seconds).
Change in UPDRS Total score (Part I-IV) [efficacy] | Week 40, Week 53 and Week 65
  Change in severity of PD non-motor and motor symptoms assessed by UPDRS Part I-IV total scores (Parts I, II and IV in ON-state; Part III in OFF-state): Part 1 (scored 0-16) Mentation, behaviour and mood. Part 2 (scored 0-52) Activities of daily living. Part 3 (scored 0-108) Motor examination. Part 4 (scored 0-23) Complications of therapy. The total score is 0-199 (0=totally healthy; 199=worst possible).
Change in home diary score [efficacy] | Weeks 40, 45, 49, 49, 53, 57, 61 and 65
  Change in functional status of the patient's dyskinesias assessed by home diary score for three-day period. Each half hour is scored: sleep, OFF, ON without dyskinesias, ON with non-troublesome dyskinesias, ON with troublesome dyskinesias. The total time in each state over 3 days is recorded (in hours). The total "bad time" is defined as "OFF time" and "ON time with troublesome dyskinesia". The total "good time" is defined as "ON time without dyskinesia" or "ON time with non-troublesome dyskinesia".
Change in PDQ-39 (Parkinson's Disease Questionnaire) score [efficacy] | Week 40, Week 53 and Week 65
  Changes in health and daily activity assessed by a self-administered PDQ-39 questionnaire comprising of 39 questions related to eight key areas of health in Parkinson's patients: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. Each question is evaluated on a scale of five terms "Never", "Occasionally", "Sometimes", "Often" or "Always or cannot do at all".
Change in CGI-I (Clinical Global Impression - Improvement) scale [efficacy] | Weeks 40, 45, 49, 53, 57, 61 and 65
  Change in mental status as measured by CGI-I scale rated by the clinical on a seven-point scale 1-7 (1=very much improved, 4=no change, 7=very much worse).
Occurrence of blockage [performance assessment] | Week 41, 45, 49, 53, 57 and Week 61
  Occurrence of blockage of implanted catheter preventing or limiting infusion assessed by measuring catheter pressure at the infusion pump during infusion (in mmHg).
Stability of transcutaneous port: Inability to start infusion due to connectivity problem in Drug Delivery System | Week 41 to Week 61
  The stability of transcutaneous port is evaluated by recording the cases when the infusion in an individual patient has not been able to start due to connectivity problem between the external infusion set and the transcutaneous port.

OTHER OUTCOMES:
Change in DAT (dopamine transporter)-PET imaging [exploratory] | Week 63
  Change in caudate and putamen DAT availability using PET imaging.
Change in alpha-synuclein levels [exploratory] | Week 40, Week Week 61 and Week 65
  Changes in serum and CSF (cerebrospinal fluid) concentrations of various α-synuclein species
Distribution of CDNF: blood serum [exploratory] | Week 61
  Concentration of CDNF in serum before and two timepoints after infusion (in ng/ml)
Distribution of CDNF: cerebrospinal fluid [exploratory] | Week 61
  Maximum concentration (Cmax) of CDNF in cerebrospinal fluid (CSF) after infusion (in ng/ml)
Change in daily activity measurement [exploratory] | Weeks 40, 45, 49, 53, 57, 61 and 65
  Change in daily activity measured by Parkinson's KinetiGraph™ (PKG™) Data Logger: dyskinesia, bradykinesia, tremor, immobility plot, fluctuation score. The PKG units are: Bradykinesia score in % from normal controls, and, Dyskinesia score in % from normal controls. The Fluctuation and Dyskinesia score (FDS) for normal controls is in the range of 7.8-12.8: a lower score indicates bradykinesia and a higher score indicates dyskinesia.
Coverage of infusate in target anatomy assessed by Magnetic resonance imaging | Week 61
  Coverage of the infusate in target anatomy assessed by MRI (Magnetic resonance imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Per Svenningsson, MD, Prof., Principal Investigator — Karolinska University Hospital
Locations (3):
- Helsinki University Hospital, Helsinki, Finland
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No